CLINICAL TRIAL: NCT03608475
Title: A Non-Inferiority Trial Assessing a Limited Ultrasound Protocol in the Treatment of Developmental Dysplasia of the Hip
Brief Title: Assessing a Limited Ultrasound Protocol in DDH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Simon Kelley, Orthopaedic Surgeon, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB1000056980
Record Dates: First submitted 2018-06-20; First posted 2018-08-01 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Developmental Dysplasia of the Hip
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive Ultrasound Group (Active Comparator): Children in the comprehensive ultrasound protocol group will follow the current standardized treatment protocol used at the Hospital for Sick Children in Toronto, Canada. For children presenting with stable hip dysplasia, Pavlik harness (PH) treatment is initiated at the initial visit (week 0) and runs for a total of 12 weeks. Children return to clinic at weeks 2, 5, 8 and 12 for clinical and ultrasound examinations to ensure that the harness is fitting correctly, to screen for PH complications and to monitor acetabular development.
  Interventions: Other: Standard Ultrasound Imaging
- Limited Ultrasound Group (Experimental): Children in the limited ultrasound protocol group will receive the same treatment as described for the comprehensive ultrasound group above, except the ultrasound imaging conducted at weeks 2, 5 and 8 will be omitted. Children will still return to clinic at 2, 5, and 8 weeks for clinical examination, which includes the assessment of the Pavlik harness fit and screening for complications.
  Interventions: Other: Limited Ultrasound Imaging

INTERVENTIONS:
Other: Limited Ultrasound Imaging — Ultrasound imaging will not be performed at the 2, 5 and 8 week clinic visits
  Arms: Limited Ultrasound Group
Other: Standard Ultrasound Imaging — Ultrasound imaging will be performed at all clinic visits
  Arms: Comprehensive Ultrasound Group

SUMMARY:
Developmental Dysplasia of the Hip (DDH) is a common diagnosis in children that if untreated may lead to degeneration and arthritis of the hip joint at a young age. Ultrasound imaging is used to monitor progress of the developing hip joint during treatment. Initial data from our practice suggests that interim ultrasounds do not alter the course or outcome of treatment. Additionally, these ultrasounds add significant time to clinic visits and carry a substantial cost to the health care system. The goal of this study is to determine if limiting the number of ultrasounds during treatment results in the same outcomes while also evaluating the amount of time and money saved by omitting the ultrasounds.

ELIGIBILITY:
Inclusion Criteria:

* Aged 0-6 months at time of diagnosis
* Clinical and Ultrasound diagnosis of stable developmental dysplasia of the hip
* Children with dislocated/ unstable DDH will be included once the hip becomes stable
* Treated with Pavlik harness
* Assessed and treated at the SickKids Baby Hip Clinic

Exclusion Criteria:

* Underlying neuromuscular disease
* Teratologic hip dysplasia
* Prior treatment at other institutions
* Non-compliance with treatment protocol

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Acetabular Index | When patient reaches 1 year of age
  Acetabular Index will be measured on a supine anteroposterior (AP) radiograph of the pelvis
International Hip Dysplasia Institute Score | When patient reaches 1 year of age
  The International Hip Dysplasia Institute (IHDI) grade will be measured from a radiograph of the pelvis. The score classifies hips into one of four groups based on the position of the proximal femoral metaphysis in relation to the acetabulum. The scores grade severity from Grade 1 as the mildest type to Grade 4 as the most severe type of hip dislocation.

SECONDARY OUTCOMES:
Complication Rate | Through study completion, an average of two years
  The frequency of complications between the treatment groups will be compared
Health Care Costs | Through study completion, an average of two years
  The difference in cost between the two treatment arms will be the cost of 3 diagnostic ultrasounds
Hospital Appointment Duration | Through study completion, an average of two years
  Calculating time between registering at Ultrasound and registering at the Orthopaedic clinic will provide a measurement of time savings in the limited ultrasound protocol group

CONTACTS AND LOCATIONS:
Overall Officials: Simon P Kelley, PhD, FRCS, Principal Investigator — The Hospital for Sick Children, Toronto, Ontario, Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No